CLINICAL TRIAL: NCT05834114
Title: The Effects of Mckenzie Protocol Versus Rhythmic Stabilization Technique on Pain, Range of Motion and Disability in Chronic Neck Pain.
Brief Title: Mckenzie and Rhythmical Stabilization Technique on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0108 Mustajab
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
Keywords: Mckenzie protocol; Rhythmic Stabilization technique
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: blinding
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie protocol (Experimental): In this group, 20 participants will be included. the interventions will be given for 15 mint. The exercises then repeated five or six times in a Session. the session will be of 45 mins, 3 session per week.
  Interventions: Other: Mckenzie protocol
- Rhythmic stabilization technique (Active Comparator): In this group, 20 participants will be included. Rhythmic Stabilization with traditional physical therapy will be given for 3 sessions of 45 minutes a week, over a period of 10 weeks.
  Interventions: Other: Rhythmic Stabilization technique

INTERVENTIONS:
Other: Mckenzie protocol — In this group 20 participants will receive McKenzie protocol with conventional physical therapy. Participants will be asked to sit to treat extension deficit. The participant will be in a comfortable sitting position with a proper back support. Head is kept in forward facing without any up and done movement (10 to 15 times). Then, he restored the neutral sitting posture, and at the end of the range of motion (ROM), he' tuck in" chin by pushing the chin with his fingers (10 to 15 times). Subsequently, the participant will be requested to return to the original position while the therapist one hand's forefinger placed alongside the participant's mandible (to stabilize the head at full retraction position), and the heel of the other hand placed on the first or second dorsal vertebra (to provide posterior-anterior force). The exercises then repeated five or six times in a Session. the session will be of 45 mins, 3 session per week.
  Other Names: McKenzie protocol for neck pain
  Arms: McKenzie protocol
Other: Rhythmic Stabilization technique — In this group participants will receive Rhythmic stabilization, with Conventional physiotherapy treatment the flexion , extension exercises performed. During flexion pattern the experimenter stood at the right side of patient and used his tip of fingers at chin. The experimenter then put his left hand at anterior side of head to apply resistance. then extension pattern is resisted and asked patient to match my resistance. The experimenter provided resistance against right rotation and lateral flexion provided during the exercise in order to induce strong muscle contractions. 3 sessions of 45 minutes a week, over a period of 10 weeks.
  Other Names: Rhythmic Stabilization technique in neck pain
  Arms: Rhythmic stabilization technique

SUMMARY:
The study will be randomized clinical trial. Total 40 subjects will be assigned randomly by using non probability convenient into two groups. Group A will be given McKenzie protocol, with conventional physiotherapy treatment while Group B is Rhythmic stabilization group who will receive rhythmic stabilization, with conventional physiotherapy. After confirmation of diagnosis with medical history and physical examination numeric pain rating scale (NPRS) and Neck disability index (NDI) would be used as an outcome measure tools for pain and disability respectively. Measure will be taken by goniometer. After data collection from defined study setting,data will be entered and analyzed at Riphah International University, Lahore.

DETAILED DESCRIPTION:
Neck pain is a very common ailment that results in a great deal of suffering, impairment, and financial expense. The International Association for the Study of Pain is defined as Pain perceived as arising from anywhere within the region bounded superiorly by superior nuchal line, inferior by an unoriginally transverse line through the tip of first thoracic spinous process, and laterally by sagittal plane tangential to the lateral border of neck. According to the study's findings, 69% of Balochistan University undergraduate students in Quetta, Pakistan, experienced neck pain. Pain in many cervical spine structures has the potential to become chronic neck pain. In epidemiologic research, pain is considered chronic if it lasts more than three months to six months, or five years.

McKenzie's treatment regimens were first used in Sweden in 1985 to address mechanical spine patient issues. For these kinds of patients, protocols were often employed in the 1990s. Repeated neck retraction exercises considerably lessen the pain and restore the cervical spine's lordosis curve in individuals with spinal pain.

Rhythmic Stabilization is characterized by isometric contractions against the resistance provided by the therapist, with the subject trying to maintain their position as the therapist changes the direction of resistance. Both techniques are effective in pain and range of motion in chronic neck pain.

McKenzie protocol and rhythmic stabilization are both studied individually before but their effects are not compared previously.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50
* Localized chronic neck pain for more than 3 months.

Exclusion Criteria:

* Participants suffering their neck pain was caused by any other complications.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | 3 weeks
  NPRS is based on 11-point numerical rating scale for determining pain intensity, 0(no pain) to 10(worst pain imaginable) pain intensity. On average over the past 2 day how bad has your pain been.
Neck disability index | 3 weeks
  The Neck Disability Index (NDI) (modification of the Oswestry Low Back Pain Disability Index).
  (0-8%) no disability, ( 10 - 28%) mild disability, (30-48% ) moderate disability, (50- 64%) severe disability, (70-100%) complete disability

SECONDARY OUTCOMES:
The Universal goniometer | 3 weeks
  It is used to measure ranges of neck flexion, extension, lateral rotation(right, left), Side bending (right, left)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Ghurki Trust Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No